CLINICAL TRIAL: NCT00689923
Title: Vertebroplasty Using Real-Time, Fluoroscopy-Controlled, Catheter-Assisted, Low-Viscosity Cement Injection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200710029R; 200710029R
Record Dates: First submitted 2008-06-01; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Osteoporosis; Compression Fracture
MeSH Terms: conditions — Osteoporosis; Fractures, Compression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Th low viscosity cement injection is safe in vertebroplasty procedure with Comparacle out come in pain relief.

DETAILED DESCRIPTION:
Pain relief; Comparatle

Cement Leakage; Comparacle

Irradiation dose：less

ELIGIBILITY:
Inclusion Criteria:

* all painful fracture that can not be relieved by pain killer.

Exclusion Criteria:

* infection and malignancy in local region

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: painful vertebral compression fracture
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
pain relief | immediately after procedure

SECONDARY OUTCOMES:
cement leak | immediate after procedure